CLINICAL TRIAL: NCT02144662
Title: To Investigate Prognostic Factors for Visual Improvement in Patients Undergoing Intravitreal Ranibizumab for Retinal Vein Occlusion
Brief Title: Prognostic Factors for Visual Improvement in Patients Undergoing Intravitreal Ranibizumab for Retinal Vein Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Marianna University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiro Kogo, Ophthalmology, St. Marianna University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STM3247
Record Dates: First submitted 2014-03-22; First posted 2014-05-22 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Researcher-Subject Relations
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab (Experimental): Ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.5mg ranibizumab intravitreal injection
  Other Names: Lucentis

SUMMARY:
Primary Objective: To investigate the pretreatment quantitative factors as shown in SD-OCT images that correlate with posttreatment VA in patients who underwent intravitreal Lucentis (Ranibizumab) for RVO.

Secondary Objectives: Correlations between posttreatment BCVA and pretreatment factors were evaluated, including age, pretreatment BCVA, photoreceptor outer segment (PROS) length, central foveal thickness (CFT), outer foveal thickness (OFT), and outer nuclear layer thickness (ONLT). The factors influencing posttreatment BCVA were evaluated using multiple regression analysis.

Detailed information on macular morphology, such as the photoreceptor IS/OS junction and ELM, can be obtained in SD-OCT. Some OCT studies evaluated other quantitative factors in eye disease. It was reported that PROS length was correlated with BCVA in patients with DME.¹ Other investigators suggested that the thickness, area, and volume of the outer layer were correlated with BCVA in patients with dry age-related macular degeneration (AMD).² Outer foveal thickness (OFT) and relative reflectivity of the outer nuclear layer (ONL) were associated with BCVA in patients with macular hole.3, 4 The volume of the ONL was found to be associated with BCVA in patients with AMD.5 The aim of this study was to investigate the pretreatment quantitative factors as shown in SD-OCT images that correlate with posttreatment VA in patients who underwent intravitreal Lucentis (Ranibizumab) for RVO.

DETAILED DESCRIPTION:
Detailed information on macular morphology, such as the photoreceptor IS/OS junction and ELM, can be obtained in SD-OCT. Some OCT studies evaluated other quantitative factors in eye disease. It was reported that PROS length was correlated with BCVA in patients with DME.¹ Other investigators suggested that the thickness, area, and volume of the outer layer were correlated with BCVA in patients with dry age-related macular degeneration (AMD).² OFT and relative reflectivity of the ONL were associated with BCVA in patients with macular hole.3, 4 The volume of the ONL was found to be associated with BCVA in patients with AMD.5 The aim of this study was to investigate the pretreatment quantitative factors as shown in SD-OCT images that correlate with posttreatment VA in patients who underwent intravitreal Lucentis (Ranibizumab) for RVO.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, Patient of RVO, BCVA ≥ 0.1 (decimal visual acuity), Mean VRT≥ 250 μm
* signed informed consent

Exclusion Criteria:

* Laser photocoagulation for ME ≤ 4 months prior to initiation of this study therapy
* Intraocular corticosteroid use ≤ 3 months prior to initiation of this study therapy
* History of anti-VEGF treatment (intravitreal ≤3 months prior to initiation of this study therapy, systemic ≤ 6 months prior to initiation of this study therapy)
* Stroke or myocardial infarction ≤ 3 months prior to initiation of this study
* Pregnancy or potential pregnancy, and breastfeeding
* Severe liver dysfunction, severe CKD/hemodialysis, uncontrolled DM (HbA1c>10), uncontrolled hypertension (BP≥ 160/100 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-01-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity at 1 year after primary treatment | 1 year

SECONDARY OUTCOMES:
age, past medical history, complication (ex. Hypertension, Hyperlipidemia etc.), pretreatment BCVA, the photoreceptor outer segment (PROS) length, central foveal thickness (CFT), outer foveal thickness (OFT), and outer nuclear layer thickness (ONLT) | baseline, 3months, 6months, 9month and 12months

CONTACTS AND LOCATIONS:
Overall Officials: Jiro Kogo, M.D., Ph. D., Principal Investigator — St. Marianna University School of Medicine